CLINICAL TRIAL: NCT00701987
Title: Dose-escalating, Pilot Study to Assess the Safety, Tolerability, and Preliminary Efficacy of ALS-357 Topically Administered to Patients With Cutaneous Metastatic Melanoma
Brief Title: Safety, Tolerability, and Preliminary Efficacy Study of ALS-357 in Patients With Cutaneous Metastatic Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Life Sciences, Inc. (Industry)
Responsible Party: David A. Eiznhamer, Executive Vice President, Clinical Development, Advanced Life Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALS-357-001
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Melanoma
Keywords: Cutaneous Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): ALS-357 applied topically twice weekly for four weeks.
  Interventions: Drug: ALS-357
- 2 (Experimental): ALS-357 applied topically every other day for four weeks.
  Interventions: Drug: ALS-357
- 3 (Experimental): ALS-357 applied topically once daily for four weeks.
  Interventions: Drug: ALS-357
- 4 (Experimental): ALS-357 applied topically twice daily for four weeks.
  Interventions: Drug: ALS-357

INTERVENTIONS:
Drug: ALS-357 — Topical application of ALS-357

SUMMARY:
A phase I trial to evaluate the safety and tolerability of ALS-357 when administered for four weeks as a topical ointment, in escalating doses, to patients with cutaneous metastatic melanoma and to evaluate the effect of escalating doses of topically applied ALS-357 on histological remission of cutaneous metastatic melanoma and induction of apoptotic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Study Participants must be 18 years or older.
* Study Participants must have 2 sites of cutaneous metastatic melanoma that can not be removed with surgery.
* Study Participants may have been previously treated with chemotherapy or immunotherapy but not with in 4 weeks of first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ALS-357 when administered for four weeks as a topical ointment, in escalating doses, to patients with cutaneous metastatic melanoma. | Day 8, 15, 22, 29 and 43
Evaluate the effect of escalating doses of topically applied ALS-357 on histological remission of cutaneous metastatic melanoma and induction of apoptotic biomarkers. | Day 8, 15, 22, 29 and 43

SECONDARY OUTCOMES:
Evaluate differences in induction of apoptosis in treated versus control lesions via TUNEL assay. | Day 15, 29 and 43
Nucleic Acid will be isolated from portions of the biopsies to be utilized for gene expression profiling by various analytical platforms and correlated with other apoptotic in situ and surface protein expression pathways. | Day 15, 29 and 43
Evaluate the plasma concentration of ALS-357 at each scheduled study visit. | Day 1, 8, 15, 22, 29 and 43

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kuzel, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States